CLINICAL TRIAL: NCT03565055
Title: From Prevention to Community Integration: Service Models, Intervention Strategies, and Outcome Evaluation for Recovery From Severe Mental Illness in Chinese Communities (Hong Kong and Beijing)
Brief Title: From Prevention to Community Integration: IPCST for Severe Mental Illness in Chinese Communities (Hong Kong and Beijing)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSANG Hector Wing-Hong, Professor and Head, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-ZVKP
Record Dates: First submitted 2017-08-28; First posted 2018-06-21 (Actual); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPCST (Experimental): Intervention = Patients that participate in IPCST programme
  Interventions: Behavioral: IPCST
- E.A.S.Y (Active Comparator): Treatment as usual = Patients of E.A.S.Y Programme in HK Kwai Chung Hospital
  Interventions: Behavioral: E.A.S.Y

INTERVENTIONS:
Behavioral: IPCST — Integrative Psychosocial & Community Skills Training (IPCST) programme
  The IPCST programme includes:
  1. psychoeducation, internalized stigma reduction, & strength and coping enhancement
  2. motivational interviewing skills
  3. Neurocognitive and social cognitive training (Au, Tsang, So, Bell, Cheung, et al., 2015)
  4. augmented supported employment with social skills training (Tsang, Fung, Li, Leung & Cheung, 2010) and
  5. family and patient involvement in care
  Arms: IPCST
Behavioral: E.A.S.Y — The E.A.S.Y. (Early Assessment Service for Young People with Early Psychosis) Programme is a service programme for people suffering from early psychosis.
  The E.A.S.Y programme includes:
  1. Extensive public education
  2. Early referral and assessment
  3. Ongoing treatment services
  Arms: E.A.S.Y

SUMMARY:
This research project aims at early detection, early intervention, and recovery of individuals with psychosis and prevention of their family members who are at high risk of having developmental problems and developing psychosis episode in later stages of their life.

It consists of two major parts with the following study designs & aims:

Part I : Developing a comprehensive and integrative psychosocial and community skills training programme (IPCST) and conducing a pilot randomised controlled trial to compare the study outcomes between the two settings in Hong Kong and Beijing.

1. To develop IPCST as an innovative intervention model targeting individuals with first or recent onset of psychosis to reduce their stay in mental hospital and bridges them to independent living in the community with optimal social and professional support;
2. To evaluate IPCST in terms of the clinical, vocational, and psychosocial outcomes of participants using a randomized controlled trial design and compare these outcomes between Hong Kong and Beijing;
3. To examine the cost-effectiveness of IPCST in the two cities; and
4. To train professionals and research personnel in Hong Kong and mainland for implementation

Part II: Exploring the health needs of younger family members of individuals with early psychosis and the strategies in preventing this clinical high risk group from developing psychotic episode and developmental problems in later stages of their lives.

1. To identify the potential developmental problems or sufferings of theses younger family members living with patients with mental illness;
2. To provide baseline assessment of their psychosocial stress, mental health, and quality of life;
3. To identify interventions that may prevent them from developing psychosis and other developmental problems and improve their mental health.

DETAILED DESCRIPTION:
This research is to develop and test on a pilot basis the clinical efficacy of the IPCST on the clinical and recovery outcomes of outpatients with first and recent-onset psychosis in one-year follow-up period in one regional outpatient care service of both Hong Kong and Beijing, China. All outcomes will be assessed by a trained Research Assistant who is blind to group assignment in each city separately. In Hong Kong, the study venue will be one Early Assessment Service for Young People with Early Psychosis (EASY) in Kwai Chung Hospital under the Kowloon West Hospital Cluster, Hospital Authority Hong Kong. In Beijing, the study venues consist of the Sixth Hospital of Peking University, the Chaoyang Third Hospital, and the Haidian Mental Health Hospital.

In both sites, the study venues are serving for first or recent-onset psychosis residing in the community.

Similar to previous psychosocial interventional studies, the primary outcomes of this study are patients' mental status and level of functioning. Secondary outcomes include the rate and length of psychiatric hospitalizations, vocational status, social skills, family functioning, and quality of life.

A total of 100 participants would be recruited for this project, 50 to be recruited from Hong Kong Kwai Chung; 50 to be recruited from mainland China sites.

Part I: Participants of this part will be randomly allocated to experimental or control group.

Experimental group participants will receive a 12-week, 48-hours of IPCST programme which includes both individual and group training on psychoeducation, motivational interviewing skills, neurocognitive and social cognition, and augmented supported employment with social skills.

Control group participants will receive the usual psychiatric treatment they have been receiving from the hospital.

All participants will receive assessment on their primary (symptom severity and functioning) and secondary (re-hospitalisation rates, family functioning, social skills, and employment status and satisfaction, and quality of life) outcomes at baseline and immediately (Post-test 1), 6 months (Post-test 2), and 12 months (Post-test 3) after completion of the interventions by a research assistant. Each assessment episode lasts about 1.5 hours.

Part II: Participants of this part will undergo a 30 minutes to 1 hour individual interview conducted by a research assistant that covers semi-structured open-ended questions and basic assessment of psychosocial stress, health and mental health status, and quality of life using quantitative measures.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong/ China residents
* Age between 18-55 years;
* Primary diagnosis of psychosis (not more than 12 months of clinical diagnosis) by psychiatrist and confirmed with the SCID-I for DSM-IV TR Axis I Disorders (Biometrics Research, 2002);
* Primary six or above education;
* Mentally competent to follow the instructions and training and give informed written consent, as suggested by the attending psychiatrist;
* Able to communicate in Chinese;
* Intend to seek employment.

Exclusion Criteria:

* Co-morbidity of learning disability, neurological disorder (e.g., epilepsy) and organic brain disease, or clinically significant medical diseases;
* Recently participated or are participating in other structured psychosocial intervention, and/or
* Visual, language or communication difficulty.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change of Positive and Negative Syndrome Scale (PANSS) score | Baseline, Completion of the 3-month program, and follow up at 6-, 12- month
  The Positive and Negative Syndrome Scale (PANSS) is a medical scale used for measuring symptom severity of patients with schizophrenia.
  Participants will be assessed by medical specialist who will complete their PANSS at baseline, immediately following the completion of the 3-month program, and at 6- & 12- months after completion of the program.
  The Change of PANSS score over the above time course is the study's primary outcome measure.
Change of The Personal and Social Performance Scale (PSP) score | Baseline, Completion of the 3-month program, and follow up at 6-, 12- month
  The Personal and Social Performance scale (PSP) is widely used to assess social functioning in patients with schizophrenia.
  Participants will be assessed by medical specialist who will complete their PSP score at baseline, immediately following the completion of the 3-month program, and at 6- & 12- months after completion of the program.
  The Change of PSP score over the above time course is the study's primary outcome measure.

SECONDARY OUTCOMES:
Change of Employment Outcome Checklist (EOC) score | Baseline, Completion of the 3-month program, and follow up at 6-, 12- month
  The Employment Outcome Checklist (EOC) is used to assess participants' employment outcomes such as the number of job interviews attended, the number of jobs obtained, number of hours per week worked, and salary received from each of the jobs that were obtained .
  Participants will be assessed by research assistant who will complete their EOC questionnaire at baseline, immediately following the completion of the 3-month program, and at 6- & 12- months after completion of the program.
  The Changes in EOC over the above time course is the study's secondary outcome measure.
Change of The Schizophrenia Quality of Life Scale Revision 4 (SQLS-R4) score | Baseline, Completion of the 3-month program, and follow up at 6-, 12- month
  The Schizophrenia Quality of Life Scale Revision 4 (SQLS-R4) is a self-report quality of life measure for people with schizophrenia.
  Participants complete on their own the SQLS-R4 questionnaire at baseline, immediately following the completion of the 3-month program, and at 6- & 12- months after completion of the program.
  The Change of SQLS-R4 score over the above time course is the study's secondary outcome measure.
Change of the Vocational Social Skills Assessment Scale (VSSS) score | Baseline, Completion of the 3-month program, and follow up at 6-, 12- month
  The Vocational Social Skills Assessment Scale (VSSS) is a self-administered checklist that measures the participants' subjective perception of their competence in handling work-related social situations.
  Participants complete on their own the VSSS questionnaire at baseline, immediately following the completion of the 3-month program, and at 6- & 12- months after completion of the program.
  The Change of VSSS score over the above time course is the study's secondary outcome measure.
Change of Re-hospitalization rate | Baseline, Completion of the 3-month program, and follow up at 6-, 12- month
  Re-Hospitalization rate measured at Baseline, Completion of the 3-month program, and follow up at 6-, 12- month
Change of outpatient follow-up rate | Baseline, Completion of the 3-month program, and follow up at 6-, 12- month
  The changes in outpatient follow-up rate measured at Baseline, Completion of the 3-month program, and follow up at 6-, 12- month